CLINICAL TRIAL: NCT05784883
Title: Prevalence, Mechanisms, and Outcome of Tricuspid Valve Regurgitation in the Elderly
Brief Title: Tricuspid Regurgitation in the ElderlY
Acronym: TREY
Status: Active, not recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohammad Abdelghani, Lecturer of Cardiology - Cardiology Consultant, Al-Azhar University
Other Study IDs: ACRI-01
Record Dates: First submitted 2023-02-25; First posted 2023-03-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-08

CONDITIONS: Tricuspid Regurgitation
Keywords: Valvular heart disease; Tricuspid regurgitation; Elderly; Geriatric; Echocardiography
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Consecutive patients ≥60-year-old presenting to the echocardiography clinic
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — A comprehensive 2- and 3-dimensional transthoracic echocardiography (TTE) assessment of the tricuspid valve and right side of the heart at baseline.

SUMMARY:
Tricuspid regurgitation (TR) is the second most common VHD after MR. Its prevalence also increases with age, with an estimated incidence of up to 6% in elderly population. When adjusted to age (among other confounders), survival is worse for patients with moderate and severe TR. We aim to explore the prevalence, mechanisms, and clinical implications of tricuspid valve regurgitation in elderly subjects screened at a tertiary center in Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All comer patients ≥60-year-old presenting to the echocardiography clinic

Exclusion Criteria:

* Poor acoustic window.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients ≥ 60 years old presenting to the echocardiography clinic.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of tricuspid valve regurgitation in the elderly | Baseline (at enrolment)
  Prevalence of mild, moderate, and severe TR in enrolled patients
All-cause mortality | At 6 months
  Incidence of death from any cause
Cardiovascular mortality | At 6 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalization for congestive heart failure | At 6 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization.

SECONDARY OUTCOMES:
Classification of tricuspid valve regurgitation in the elderly | Baseline
  Classify the type of TR according to the main morphologic and/or functional abnormality. The classification will be done according to the following proposal, the TR could be 1- primary (organic) if there is an anatomical abnormality of the tricuspid valve apparatus. 2- secondary (functional) if the tricuspid valve apparatus was normal but the TR due to annular dilation. If the annular dilation is due to right ventricular volume or/and pressure overload, the TR will classify as ventricular TR, whereas if the annular dilation is due to atrial fibrillation, the TR will classify as atrial TR. The last type of TR is due to the implantation of a cardiac implantable electronic device (CIED) which will classify as CIED-related TR.
Change in New York Heart Association (NYHA) functional class | At 6, 12 and 60 months
  New York Heart Association [NYHA] functional class (I-IV) will be assessed in all participants at baseline and at follow-up visits (or by phone interviews).
  NYHA Class I: No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  NYHA Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  NYHA Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  NYHA Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
All-cause mortality | At 12 and 60 months
  Incidence of death from any cause
Cardiovascular mortality | At 12 and 60 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalization for congestive heart failure | At 12 and 60 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Abdelghani, MD, PhD, Principal Investigator — Al-Azhar Cardiology Research Institute
Locations (1):
- Al Hussein University Hospital of Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelghani M, Mohey S, Elnahas AM, Elshernouby KA, Muharram M, Gebaly M, Mokhaimar B, Elbadawi M, Diab RA, Abdelshafy M, Soliman O, Attia W. Tricuspid valve and right-heart chamber remodelling in elderly subjects with secondary tricuspid regurgitation. Acta Cardiol. 2024 Nov;79(9):1011-1020. doi: 10.1080/00015385.2024.2359657. Epub 2024 May 31. PMID 38818766